CLINICAL TRIAL: NCT01212796
Title: Second and Further Allogeneic Stem Cell Transplantation Following Relapse After Allogeneic Transplant in Haematological Malignancies: Retrospective Results of the GETH
Brief Title: Allo After Allo Stem Cell Transplantation Following Relapse After Allogeneic Transplant in Haematological Malignancies: Retrospective Results of the GETH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Grupo Espanol de trasplantes hematopoyeticos y terapia celular (Other)
Responsible Party: Angel Cedillo, GETH
Other Study IDs: GET-ALO-2010-01; get-alo-2010-01
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Allogeneic Stem Cell Transplantation
Keywords: allogeneic stem cell transplantation

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The allogeneic hematopoietic stem cell marrow is the only curative treatment for many hematologic malignancies. However, many patients relapse in these situations to be therapeutic possibilities scarce and mixed. Chemotherapy in these situations does not show good results and new drugs have not yet demonstrated the effectiveness desired.

Another therapeutic approach after relapse post allogeneic transplant is to resubmit the allogeneic transplant patient to patient. In this clinical situation is little known. All previous studies are retrospective, the data provided are of little statistical value and heterogeneous patient samples.

The GETH (Grupo Espanol de trasplantes hematopoyeticos y terapia celular) has included in its database a figure around 350 seconds allogeneic transplants. Comparing this with the studies published so far, this would be the largest retrospective series published size compared to second allogeneic transplants.

DETAILED DESCRIPTION:
It reviewed 350 patients who underwent allogeneic 2 or more between the beginning of monitoring and the end of 2009, end of follow-up. Is a multicenter study of row should include all possible patients who take the appropriate data. To all centers contributing patients to the study, were asked to fill out basic information related to the data sheets of the EBMT report (MED-A and MED-B).

To collect these forms of EBMT, patients have previously authorized through the informed consent of this information collection.

It will include basic descriptive characteristics of the cohort and comparisons between groups were conducted to check if the sample is homogeneous.

The analysis is divided into descriptive data collection related to the transplant, both prior to transplantation and on during it. It also collected data related to transplant once done this.

FINDINGS AND PURPOSE The main variables to be analyzed are: overall survival, disease-free survival and progression, relapse rate and transplant-related mortality.

Secondary endpoints to be analyzed can vary once made the data collection. Yet between them will include: incidence of graft-versus-host disease (both acute and chronic), incidence of infections.

The purpose of this study is the description of variables that can predict the success or failure of making a second allogeneic transplant after the first relapse. These variables were also analyzed for third or subsequent transplants.

Also seeks to differentiate risk groups among patients. The novelty of this study could provide regarding previously published studies is the description of third or subsequent transplants, so far there are few references to this in the literature to date.

FINANCING This study does not require funding.

CONFLICT OF INTEREST There is no conflict of interest

DATA COLLECTION PERIOD AEMET submission and acceptance: 1-2 months. Aceppt (SEPT-10-2010) Data collection: 3 - 6 months Results: at 6 - 9 months Publication and presentation at conferences, at 12 months

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent 2 or more allogeneic transplants and the beginning of monitoring and the end of 2009, end of follow-up.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent 2 or more allogeneic transplants in Spanish hospitals between the beginning of monitoring and the end of 2009, end of follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-03 (Estimated); Study Completion 2011-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Duarte R Palomino, MD, Principal Investigator — Grupo Espanol de trasplantes hematopoyeticos y terapia celular